CLINICAL TRIAL: NCT06668974
Title: Bidirectional Mendelian Randomization Study Reveals Causal Associations Between Allergic Rhinitis and Asthma
Brief Title: Causal Associations Between Allergic Rhinitis and Asthma
Status: Completed | Type: Observational
Sponsor: Zhibin Xu (Other)
Responsible Party: Sponsor-Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: GS-002
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: Mendelian Randomization; Genetic Association; Bidirectional Causality; Genome-Wide Association Study (GWAS); Respiratory Diseases
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Respiratory Tract Diseases | interventions — Mendelian Randomization Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allergic Rhinitis Cohort: This cohort consists of individuals with allergic rhinitis and a control group from the UK Biobank database, including 18,934 cases of allergic rhinitis and 64,595 controls. Genetic data were used to explore causal relationships with asthma.
  Interventions: Other: Mendelian Randomization
- Asthma Cohort: This cohort includes individuals with asthma and a control group from the Finnish biobank database, consisting of 20,629 cases of asthma and 135,449 controls. Genetic data were analyzed to examine causal associations with allergic rhinitis.
  Interventions: Other: Mendelian Randomization

INTERVENTIONS:
Other: Mendelian Randomization — This study utilizes a bidirectional Mendelian randomization approach to analyze genetic data from individuals with allergic rhinitis and asthma. No active intervention is applied; genetic variants serve as instrumental variables to assess causal associations between the conditions.

SUMMARY:
This study investigates the causal relationship between allergic rhinitis and asthma using a bidirectional two-sample Mendelian randomization approach. Genetic data were derived from UK Biobank for allergic rhinitis and from Finnish biobank for asthma. This analysis aims to clarify the potential causal link between these two conditions.

DETAILED DESCRIPTION:
This observational study utilizes a bidirectional two-sample Mendelian randomization (MR) analysis to examine the causal association between allergic rhinitis and asthma. The genetic data for allergic rhinitis were obtained from the UK Biobank, encompassing 18,934 cases and 64,595 controls, while asthma data were derived from a Finnish biobank, including 20,629 cases and 135,449 controls. The Mendelian randomization analysis was performed using inverse-variance weighting (IVW), Mendelian randomization-Egger (MR-Egger), and weighted median methods to ensure robust causal inference. Additional tests, such as Cochrane's Q test and Mendelian randomization pleiotropy residual sum and outlier (MR-PRESSO), were applied to assess heterogeneity and pleiotropy, enhancing the reliability of the findings. The results are expected to provide insights into the bidirectional causal relationship between allergic rhinitis and asthma, potentially informing future prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with allergic rhinitis or asthma.
* Availability of genetic data in the UK Biobank or Finnish biobank.

Exclusion Criteria:

* Individuals without genetic data.
* Participants with incomplete phenotype or genotype data.

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study includes individuals diagnosed with allergic rhinitis or asthma from the UK Biobank and Finnish biobank databases.
Sampling Method: Non-Probability Sample
Enrollment: 239607 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Causal Effect of Allergic Rhinitis on Asthma Risk | Oct 24 2024
  Estimate the causal effect of allergic rhinitis on asthma risk using bidirectional Mendelian randomization. This measure includes odds ratios (OR) derived from inverse-variance weighting (IVW), Mendelian randomization-Egger (MR-Egger), and weighted median methods.
Causal Effect of Asthma on Allergic Rhinitis Risk | Oct 24 2024
  Estimate the causal effect of asthma on allergic rhinitis risk using bidirectional Mendelian randomization. This measure includes odds ratios (OR) derived from inverse-variance weighting (IVW), Mendelian randomization-Egger (MR-Egger), and weighted median methods.

SECONDARY OUTCOMES:
Sensitivity Analysis Using MR-Egger Intercept Test | Oct 24 2024
  Perform sensitivity analysis using the Mendelian randomization-Egger (MR-Egger) intercept test to assess horizontal pleiotropy in the causal estimates between allergic rhinitis and asthma.
Sensitivity Analysis Using Leave-One-Out Test | Oct 24 2024
  Conduct a leave-one-out test to evaluate the robustness of the causal estimates between allergic rhinitis and asthma by sequentially removing each single nucleotide polymorphism (SNP).
Sensitivity Analysis Using MR-PRESSO | Oct 24 2024
  Use the Mendelian randomization pleiotropy residual sum and outlier (MR-PRESSO) test to detect and correct for outliers, assessing heterogeneity in the causal estimates between allergic rhinitis and asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Diseases, the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided